CLINICAL TRIAL: NCT02684578
Title: METforMIN: Metformin Administration for the Minimization of Geographic Atrophy Progression in Patients With Age-related Macular Degeneration
Brief Title: Metformin for the Minimization of Geographic Atrophy Progression in Patients With AMD
Acronym: METforMIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency); VA Palo Alto Health Care System (U.S. Federal Agency); University of California, Davis (Other); University of California, San Diego (Other); Northwestern University (Other); University of Illinois at Chicago (Other); Retinal Consultants Medical Group (Other); Retina Health Center (Industry); California Retina Consultants (Other); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-18258
Record Dates: First submitted 2016-02-09; First posted 2016-02-18 (Estimated); Results first posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Age-Related Macular Degeneration; Macular Degeneration, Age-Related; Dry Macular Degeneration; Geographic Atrophy
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy | interventions — Metformin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Metformin (Experimental): This arm will be receiving the study drug, Metformin, for the duration of the 24 month study. They will begin this drug on a low dose of Metformin, increasing the dosage in a step-wise fashion to avoid unwanted gastrointestinal discomfort, a common side effect when patients begin taking Metformin. During the 24 month study, subjects assigned to this arm will have 4 follow-up exams after the initial enrollment exam, at 6 month intervals.
  Interventions: Drug: Metformin
- Observe (No Intervention): This arm will maintain standard of care for dry AMD, which is observation. During the 24 month study, subjects assigned to this arm will have 4 follow-up exams after the initial enrollment exam, at 6 month intervals.

INTERVENTIONS:
Drug: Metformin
  Other Names: Glucophage
  Arms: Metformin

SUMMARY:
The purpose of this study is to determine whether metformin, an FDA-approved drug for the treatment of type II diabetes, is a safe and effective treatment to decrease the progression of geographic atrophy in non-diabetic patients with Age-related Macular Degeneration (AMD).

DETAILED DESCRIPTION:
This is a phase II, single-blind, randomized, evaluation of the safety and efficacy of metformin use to decrease geographic atrophy (GA) progression in non-diabetic patients with dry Age-related Macular Degeneration (AMD). Approximately 186 study subjects throughout four separate study sites will be randomized in a 1:1 ratio to the treatment group and the observation group. The treatment group will be assigned to the study intervention (oral Metformin) for 18 months while the observation group will receive no intervention for 18 months, instead continuing with standard of care ophthalmic exams and close monitoring of their disease. There will be one additional follow up visit at 24 months. Throughout the 24 month study period, the progression of subjects' GA or drusen growth will be measured via ocular imaging taken at standard of care follow-up examinations, including fundus autofluorescence imaging, optical coherence tomography (OCT), and fundus photography.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be >/= 55 years of age
* Subject must have evidence of advanced dry AMD, defined by the characteristic presence of drusen and/or pigmentary changes as well as geographic atrophy
* Subject must have clear ocular media and adequate pupillary dilation
* Subject must be able to swallow capsules
* Study eye must have best corrected visual acuity (BCVA) of 20/20-20/400
* Subject must be willing and able to pay for monthly prescription of Metformin HCl for 18 months in the event that their insurance carrier will not cover the cost of the drug

Exclusion Criteria:

* Subjects with insufficient baseline size of geographic atrophy, less than 1.25 mm2 (0.5 Macular Photocoagulation Study Disc Areas). GA is defined as one or more well-defined and often circular patches of partial or complete depigmentation of the RPE, typically with exposure of underlying choroidal blood vessels. Even if much of the RPE appears to be preserved and large choroidal vessels are not visible, a round patch of RPE partial depigmentation may be classified as early GA. The GA in the study eye must be able to be photographed in its entirety, and it must not be contiguous with any areas of peripapillary atrophy, which can complicate area measurements.
* Subjects who are already taking metformin for another purpose
* Subjects with type 1 or 2 diabetes
* Subjects with compromised kidney function:
* Serum creatinine ≥1.5 mg/dL for males and ≥1.4 mg/dL for females
* Subjects with moderate to severe heart failure (Class III or IV, New York Heart Association Functional Classifications)
* Subjects with Child's class C cirrhosis
* Evidence of retinal atrophy due to causes other than atrophic AMD.
* Subjects who have had anti-VEGF injections or active choroidal neovascularization in the study eye during the last 12 months
* Current evidence or history of ocular disorders in the study eye that in the opinion of the investigator confounds study outcome measures, including (but not limited to):

  1. Non-proliferative diabetic retinopathy involving 10 or more hemorrhages or microaneurysms, or active proliferative diabetic retinopathy
  2. Branch or central retinal vein or artery occlusion
  3. Macular hole
  4. Pathologic myopia
  5. Uveitis
  6. Pseudovitelliform maculopathy
  7. Intraoperative surgery within the last 90 days prior to study eye enrollment

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-04; Primary Completion 2022-04 (Actual); Study Completion 2022-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay M Stewart, MD, Principal Investigator — University of California, San Francisco
Locations (12):
- United States (12):
  - University of California, Davis, Davis, California
  - Palo Alto Veteran Affairs Medical Center, Palo Alto, California
  - Retinal Consultants Medical Group, Sacramento, California
  - San Francisco Veteran Affairs Medical Center, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - California Retina Consultants, Santa Maria, California
  - North Bay Vitreoretinal Consultants, Santa Rosa, California
  - Retina Health Center, Fort Myers, Florida
  - Northwestern University, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Oregon Health and Science University, Portland, Oregon
  - Austin Retina Associates, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Groups:
- Metformin: This arm will be receiving the study drug, Metformin, for the duration of the 24 month study. They will begin this drug on a low dose of Metformin, increasing the dosage in a step-wise fashion to avoid unwanted gastrointestinal discomfort, a common side effect when patients begin taking Metformin. During the 24 month study, subjects assigned to this arm will have 4 follow-up exams after the initial enrollment exam, at 6 month intervals.
  Metformin
- Observation: This arm will maintain standard of care for dry AMD, which is observation. During the 24 month study, subjects assigned to this arm will have 4 follow-up exams after the initial enrollment exam, at 6 month intervals.
Period: Overall Study
Arm/Group | Metformin | Observation
Started | 32; 53 eyes | 34; 57 eyes
Completed | 21; 34 eyes | 23; 37 eyes
Not Completed | 11; 19 eyes | 11; 20 eyes
Not completed — Withdrawal by Subject | 10 | 7
Not completed — Lost to Follow-up | 0 | 3
Not completed — Ineligible after reviewing baseline imaging | 1 | 0
Not completed — Missing follow-up data | 0 | 1

BASELINE CHARACTERISTICS:
Units Other Than Participants: eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Observe | Total
Number analyzed (Participants) | 32 | 34 | 66
Number analyzed (eyes) | 53 | 57 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.5 (10.9) | 79.3 (7.3) | 78.9 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 13 | 15 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 29 | 30 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 32 | 34 | 66
Presence of GA in both eyes [Count of Participants; unit: Participants] | 27 | 32 | 59
History of cardiovascular diseases [Count of Participants; unit: Participants] | 19 | 22 | 41
History of respiratory diseases [Count of Participants; unit: Participants] | 6 | 10 | 16
History of hepatobiliary diseases [Count of Participants; unit: Participants] | 1 | 3 | 4
History of gastrointestinal diseases [Count of Participants; unit: Participants] | 7 | 11 | 18
History of genitourinary diseases [Count of Participants; unit: Participants] | 5 | 9 | 14
History of endocrine diseases [Count of Participants; unit: Participants] | 5 | 6 | 11
History of hematological diseases [Count of Participants; unit: Participants] | 1 | 4 | 5
History of musculoskeletal diseases [Count of Participants; unit: Participants] | 16 | 12 | 28
History of neoplasia [Count of Participants; unit: Participants] | 4 | 4 | 8
History of neurological diseases [Count of Participants; unit: Participants] | 5 | 7 | 12
History of psychological diseases [Count of Participants; unit: Participants] | 5 | 2 | 7
History of immunological diseases [Count of Participants; unit: Participants] | 1 | 3 | 4
History of dermatological diseases [Count of Participants; unit: Participants] | 2 | 7 | 9
History of allergies [Count of Participants; unit: Participants] | 9 | 11 | 20
History of ear, nose throat diseases [Count of Participants; unit: Participants] | 7 | 5 | 12
History of other diseases [Count of Participants; unit: Participants] | 1 | 1 | 2
Number of eligible eyes [Number; unit: eyes] | 53 | 57 | 110
Best corrected visual acuity [Mean (Standard Deviation); unit: number of letters read on ETDRS] — Best corrected visual acuity (BCVA) is the best possible vision that an eye can achieve with corrective lenses (e.g., glasses or contact lenses). For this study, BCVA was measured using the Early Treatment of Diabetic Retinopathy Study (ETDRS) visual acuity charts.
  number of letters read on ETDRS | 58.5 (18.5) | 57.0 (19.4) | 57.7 (18.9)
Low luminance visual acuity [Mean (Standard Deviation); unit: number of letters read on ETDRS] — Low luminance visual acuity (LLVA) involves standard BCVA testing under low-light conditions, which is achieved by adding a neutral density filter in front of the eye. For this study, LLVA was measured using the ETDRS visual acuity charts.
  number of letters read on ETDRS | 42.8 (16.4) | 40.0 (17.9) | 41.3 (17.2)
Geographic atrophy (GA) area [Mean (Standard Deviation); unit: mm^2] — Geographic atrophy (GA) is the advanced stage of non-neovascular age-related macular degeneration (AMD). Total area of the GA lesions on fundus autofluorescence (FAF) imaging was measured using Heidelberg Eye Explorer software.
  mm^2 | 6.2 (4.4) | 8.7 (6.1) | 7.5 (5.5)
Multifocal lesion [Number; unit: eyes] | 34 | 33 | 67
Foveal center point involvement [Number; unit: eyes] | 45 | 48 | 93
Fundus autofluorescence (FAF) Pattern, "None" or "Focal" [Number; unit: eyes] — FAF pattern refers to the morphology of the GA lesion border as seen on FAF imaging. "None" indicates no or very limited increase in autofluorescence at and beyond the border of GA. "Focal" indicates GA with one or more small spots of increased autofluorescence directly adjacent to its margin. One of 3 pairs of trained, masked graders independently and manually graded FAF patterns.
  eyes | 38 | 34 | 72

OUTCOME MEASURES:

1. Primary Outcome: Fundus Autofluorescence Imaging to Measure the Rate of Change in Area of Geographic Atrophy
Description: The primary efficacy endpoint was the annualized growth rate of the square root of geographic atrophy (GA) area in mm/year in the study eye as imaged by fundus autofluorescence (FAF) imaging. Change = (Month 18 GA Area - Baseline GA Area).
Time Frame: 0 months, 18 months
Measure: Mean (Standard Deviation); unit: mm/year
Units Other Than Participants: eyes
Arm/Group | Metformin | Observation
Number analyzed (Participants) | 21 | 23
Number analyzed (eyes) | 34 | 37
mm/year | 0.41 (0.05) | 0.35 (0.05)
Statistical Analysis 1: Comparison: Metformin vs Observation; Test type: Superiority; p = 0.39, Linear mixed-effects regression — The threshold for statistical significance was p = 0.05

2. Secondary Outcome: Change in Best Corrected Visual Acuity (BCVA)
Description: BCVA is the best possible vision an eye can see with corrective lenses and is measured as then number of letters read on the ETDRS chart. Change = (Month 18 Score - Baseline Score).
Time Frame: 0 months, 18 months
Measure: Mean (Standard Error); unit: letters correctly read
Arm/Group | Metformin | Observation
Number analyzed (Participants) | 21 | 23
letters correctly read | -3.2 (0.9) | -3.2 (1.3)
Statistical Analysis 1: Comparison: Metformin vs Observation; Test type: Superiority; p = 0.97, Linear mixed-effects — The threshold for statistical significance was p = 0.05

3. Secondary Outcome: Change in Low-luminance Visual Acuity (LLVA)
Description: LLVA involves standard BCVA testing in low-light conditions, which is achieved by adding a neutral density filter in front of the eye being tested. LLVA is measured as the number of letters read on the ETDRS chart. This measure has been shown to correlate well with enlargement of GA. Change = (Month 18 Score - Baseline Score).
Time Frame: 0 months, 18 months
Measure: Mean (Standard Error); unit: letters correctly read
Arm/Group | Metformin | Observation
Number analyzed (Participants) | 21 | 23
letters correctly read | -2.1 (2.0) | -6.3 (1.9)
Statistical Analysis 1: Comparison: Metformin vs Observation; Test type: Superiority; p = 0.12, Linear mixed-effects — The threshold for statistical significance was p = 0.05

4. Secondary Outcome: Ocular Safety as Measured by the Presence of Novel Intraocular Inflammation Judged by the Investigator to be Due to the Study Drug Metformin
Description: Subjects assigned to the Metformin study arm will be assessed at each follow-up eye exam to confirm ocular safety of metformin. The Data Safety and Management Board for this study will also assess the safety of metformin at different time points throughout the study. They will formally meet to discuss study subject safety at 25% enrollment and 75% enrollment. The potential for ocular side effects due to metformin is thought to be very low, due to the large number of diabetic patients who take this drug and are followed closely for diabetic retinopathy or other ocular disease.
  This outcome measures the number of treatment arm patients who experienced adverse ocular events during 1 or more follow-up visits.
Time Frame: 0 months, 6 months, 12 months, 18 months, 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin
Number analyzed (Participants) | 21
Participants | 0

5. Secondary Outcome: Systemic Safety as Measured by Presence of Side Effects Listed on Metformin Drug Label as "Severe"
Description: These include:
  Infrequent side effects of metformin (severe):
  * Trouble Breathing
  Rare side effects of metformin (severe):
  * Increased Blood Acidity due to High Levels of Lactic Acid (Lactic acidosis)
  * Low Blood Sugar
  * Megaloblastic Anemia
  * Reaction due to an Allergy
  Subjects assigned to the Metformin study arm will be assessed for these side-effects at each follow-up eye exam to confirm ocular safety of metformin. The Data Safety and Management Board for this study will also assess the safety of metformin at different time points throughout the study. They will formally meet to discuss study subject safety at 25% enrollment and 75% enrollment.
  This outcome measures the number of treatment arm patients who experienced side effects listed on Metformin drug label as "severe" during 1 or more follow-up visits.
Time Frame: 0 months, 6 months, 12 months, 18 months, 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin
Number analyzed (Participants) | 21
Participants | 0

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Metformin | Observation
All-Cause Mortality (participants affected / at risk) | 0/32 | 2/34
Serious Adverse Events (participants affected / at risk) | 5/32 | 3/34
Other Adverse Events (participants affected / at risk) | 16/32 | 4/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=32) | Observation (N=34)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (2)
Ascending thoracic aortic aneurysm without rupture (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infectious or inflammatory pancolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=32) | Observation (N=34)
Gastrointestinal discomfort (Gastrointestinal disorders) | 5 (5) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Chest pain (General disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Fall due to dizziness (General disorders) | 1 (1) | 0 (0)
Nausea (General disorders) | 1 (1) | 1 (2)
Rash on back and abdomen (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dry eyes (Eye disorders) | 0 (0) | 1 (1)
Development of choroidal neovascularization (Eye disorders) | 0 (0) | 2 (2)
Development of subretinal hemorrhage (Eye disorders) | 1 (1) | 1 (1)
Common cold (General disorders) | 1 (1) | 0 (0)
Cough (General disorders) | 1 (1) | 0 (0)
Subjective complaint of elevated blood pressure (General disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritability and anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Heartburn (General disorders) | 1 (1) | 0 (0)
Increased lipase (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatic fibrosis of unknown origin (Hepatobiliary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT02684578/Prot_SAP_000.pdf